CLINICAL TRIAL: NCT05813951
Title: Efficacy and Safety of Continuous Versus Intermittent Linezolid Infusion in Critically Ill Patients With Septic Shock
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ibrahim Elsayed, principle investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU R235/2022
Record Dates: First submitted 2023-02-14; First posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Treatment Efficacy
MeSH Terms: interventions — Linezolid

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled study
Who Masked: Participant, Care Provider
Masking Description: . At the beginning of the study, simple randomization will be used to assign patients using the random numbers set offered by the ICU coordinator. Each patient will be assigned a randomized code consisting of two letters that indicate the intensive care unit and two digits indicating the randomization sequence.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- continuous infusion (Active Comparator): seventy Patients in the continuous infusion group will receive an intravenous loading dose of 600 mg of Linezolid for 60 min, followed by a continuous infusion of 1200 mg/day (50 mg/h)
  Interventions: Drug: Linezolid
- intermittent infusion (Active Comparator): seventy patients in the intermittent infusion group will administrate 600 mg of linezolid IV every 12 h for 60 min
  Interventions: Drug: Linezolid

INTERVENTIONS:
Drug: Linezolid — linezolid either continues infusion or standard intermittent dose
  Other Names: zyvox

SUMMARY:
The aim of study is this to evaluate the efficacy and safety of continuous linezolid infusion versus the standard regimen in treating critically ill patients with septic shock in the ICU

DETAILED DESCRIPTION:
it is Prospective randomized controlled study on One hundred forty patients to evaluate the efficacy and safety of continuous linezolid infusion versus the standard regimen in treating critically ill patients with septic shock in the ICU, Initially, each patient will be evaluated for septic shock based on the clinical criteria. Baseline microbiologic specimens will be obtained for all recruited patients through the day of diagnosis including blood C&S. Then, empirical treatment with antibiotics according to expected source of sepsis. Patients with Gram-positive cultures sensitive to Linezolid will be randomly allocated to receive Linezolid in the continuous infusion group (Group A) or conventional intermittent infusion group (Group B) in a 1:1 ratio.

Group A: seventy Patients in the continuous infusion group will receive an intravenous loading dose of 600 mg for 60 min, followed by a continuous infusion of 1200 mg/day (50 mg/h).

Group B: seventy patients in the intermittent infusion group will administrate 600 mg of linezolid IV every 12 h for 60 min.

The treatment period will be 8-10 days in both groups but might decrease or increase based on the patients' clinical response. At the beginning of the study, simple randomization will be used to assign patients using the random numbers set offered by the ICU coordinator. Each patient will be assigned a randomized code consisting of two letters that indicate the intensive care unit and two digits indicating the randomization sequence.

The end point of the study is occurrence of thrombocytopenia (decrease in platelet count ≥ 50% from baseline or a decrease in platelet count ≤ 100 × 103/mm3).

ELIGIBILITY:
Inclusion Criteria:

* adult patients aged > 18 years old
* diagnosis of septic shock (patient with septic shock can be clinically identified by a vasopressor requirement to maintain a mean arterial blood pressure of 65 mm Hg or greater and serum lactate level greater than 2 mmol\L (>18 mg\dL) in the absence of hypovolemia).
* positive culture confirming linezolid susceptibility.

Exclusion Criteria:

* Patient refusal.
* Known allergy to linezolid.
* Pregnancy and lactation.
* Severe hepatic failure (Child-Pugh C).
* Thrombocytopenia (platelet count < 80,000/mm3).
* Disseminated intravascular coagulation (DIC).
* Hematologic disease, and concurrent use of other medications that may interact with linezolid (i.e., macrolides, serotonin modulators), or drug-associated thrombocytopenia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-12-02 (Actual); Primary Completion 2023-12-02 (Estimated); Study Completion 2023-12-02 (Estimated)

PRIMARY OUTCOMES:
occurrence of medical cure | 7 days
  primary outcome defined as occurrence of medical cure on day 7 following linezolid initiation. Clinical cure will be indicated as normal body temperature(36.1 C- 37.2C).

SECONDARY OUTCOMES:
secondary outcomes | 30 days
  1. ICU stay(days)
  2. duration of hospital stay (days).
  3. duration of linezolid treatment until clinical cure(days).
  4. Mortality at the end of treatment, and 30-day mortality.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No